CLINICAL TRIAL: NCT02834364
Title: LGX818 in Combination With MEK162 in Refractory or Relapsed Multiple Myeloma Patients With BRAFV600E or BRAFV600K Mutation
Brief Title: BRAF/MEK Inhibition in Relapsed/Refractory Multiple Myeloma (BIRMA)
Acronym: GMMG-BIRMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Heidelberg Medical Center (Other)
Collaborators: Array BioPharma (Industry); German Cancer Research Center (Other); Coordinating Centre for Clinical Trials Heidelberg (Unknown); University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Marc Raab, PD Dr. med, University of Heidelberg Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLGX818ADE01T; 2014-004597-42 (EudraCT Number)
Record Dates: First submitted 2016-06-13; First posted 2016-07-15 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Relapsed or Refractory Multiple Myeloma; Patients With BRAFV600 E or BRAFV600K Mutation
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — encorafenib; binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm (Experimental): Encorafenib 450 mg. p.o.once daily and Binimetinib 45 mg p.o. twice daily until disease progression or toxicity requiring discontinuation of treatment. 1 cycle is defined as 28 days.
  Interventions: Drug: Encorafenib; Drug: Binimetinib

INTERVENTIONS:
Drug: Encorafenib — 450 mg p.o. once daily. One cycle is defined as 28 days
  Other Names: LGX818
Drug: Binimetinib — 45 mg p.o. twice daily. One cycle is defined as 28 days
  Other Names: MEK162

SUMMARY:
Trial for patients with refractory multiple myeloma after failure of at least two treatment regimens and with BRAFV600E/K Mutation to evaluate the efficacy of the kinase inhibitors Encorafenib (LGX818 in) combination with Binimetinib (MEK162).

DETAILED DESCRIPTION:
An open-label, single-arm, multi-centre phase II trial for patients with refractory multiple myeloma and with BRAFV600E/K Mutation to evaluate the efficacy of the kinase inhibitors Encorafenib (LGX818 in) combination with Binimetinib (MEK162). The patients must have received at least two prior therapy regimen (at least one immunomodulatory drug and one proteasome inhibitor).

The subjects receive LGX 818 450 mg. p.o. once daily and MEK 162 45 mg p.o. twice daily until disease progression or toxicity requiring discontinuation of treatment. 1 cycle is defined as 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has provided a signed study Informed Consent Form prior to any study-specific procedure and is able to comply with protocol requirements
2. Patients with multiple myeloma,relapsed or refractory after failure of two or more lines of systemic treatments. All patients must have received at least one immunomodulatory drug (IMiD) and a proteasome inhibitor.

   Multiple myeloma requiring systemic therapy must have been confirmed in the medical history of the patients with criteria established by the International Myeloma Working Group (IMWG) (Rajkumar V et al. Lancet International Myeloma Working Group updated criteria for the diagnosis of multiple myeloma. Lancet 2014; 15: 538-548)
3. Written confirmation of BRAFV600E mutation or BRAFV600K mutation in in the majority of myeloma cells, defined by positive IHC staining with mutations specific antibody of ≥ 50% in the respective biopsy, confirmed by DNA sequencing of the corresponding codon
4. Measurable disease, as defined as: Measurable levels of myeloma paraprotein in serum (≥ 0.5 g/dL) or urine (≥ 0.2 g/24 hours) or FLC of involved light chain > 100mg/l and abnormal FLC-ratio
5. Age ≥18
6. WHO performance status 0-3 (WHO 3 is allowed only when caused by MM and not by comorbid conditions) (see Appendix 3)
7. Negative pregnancy test within 72 hours of inclusion (women of childbearing potential): For all men and women of childbearing potential: patients must be willing and capable to use adequate contraception during the complete therapy (see also exclusion criteria).
8. All patients must agree to abstain from donating blood while on study
9. Adequate cardiac function: left ventricular ejection fraction (LVEF) ≥ 50% as determined by an echocardiogram, QTc interval ≤ 450 ms
10. Ability of subject to take oral medications
11. Ability of subject to understand character and individual consequences of clinical trial

Exclusion Criteria:

1. Patient with prior treatment with MEK and/or RAF inhibitors
2. Systemic AL amyloidosis (except for patients with AL amyloidosis of the skin or the bone marrow)
3. Patients with meningeosis or central nervous system lesion(s) caused by multiple myeloma. However, patients treated with stereotactic radiotherapy or surgery are eligible if patient remained without evidence of CNS disease progression ≥ 4 weeks.
4. History or current evidence of retinal vein occlusion (RVO) or predisposing factors to RVO (e.g. uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes)
5. History of retinal degenerative disease
6. Plasma cell leukaemia which requires the presence of 20% of plasma cell in peripheral blood leukocytes and at least 2/nl.
7. Patient has received radiotherapy (including therapeutic radioisotopes) ≤ 21 days, if not restricted to a single osteolytic lesion, or has not recovered from side effects of such therapy.
8. Patient has had major surgery within 21 days prior to starting study drug or has not recovered from major side effects of the surgery. Kyphoplasty as prevention of skeletal related events is allowed.
9. Patient is concurrently using other approved antineoplastic or any investigational agents in the last 14 days prior to start of treatment. Note: patients may have received a cumulative dose of up to 160 mg of dexamethasone or equivalent as emergency therapy within 4 weeks prior to study entry.
10. Impaired cardiovascular function or clinical significant cardiovascular disease including any of the following: Symptomatic chronic heart failure, history or current evidence of clinically significant cardiac arrhythmia and/or conduction abnormality <6 months prior to Screening except atrial fibrillation and paroxysmal supraventricular tachycardia;

    1. LVEF < 50% as determined by ECHO, or uncontrolled hypertension despite medical treatment (please refer to WHO ISH guidelines)
    2. Clinically significant resting bradycardia, unstable angina pectoris ≤ 3 months prior to starting study drug, history of acute coronary syndromes (including myocardial infarction, coronary artery bypass grafting, coronary angioplasty, or stenting) <6 months prior to screening
    3. QTcF > 450 msec
    4. patients with acute diffuse infiltrative pulmonary and pericardial disease
11. Significant hepatic dysfunction (serum bilirubin ≥ 2 mg/dl or ASAT and/or ALAT ≥ 2.5 times normal level), unless related to myeloma
12. Active hepatitis B, and/or active hepatitis C infection
13. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral LGX818/MEK162 (e.g., ulcerative diseases, uncontrolled nausea,vomiting, diarrhea, malabsorption syndrome, small bowel resection).
14. Gilbert´s syndrome
15. Patients who have neuromuscular disorders that are associated with elevated CK (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
16. Patients who are planning on embarking on a new strenuous exercise regimen after first dose of study treatment. Note: Muscular activities, such as strenuous exercise, that can result in significant increases in plasma CK levels should be avoided while on MEK162 treatment
17. Patients known to be HIV-positive
18. Patients with active, uncontrolled infections (patients successful treated with antimicrobial therapy may be enrolled at the discretion of the investigator).
19. Patient is receiving chronic treatment with systemic steroids or another immuno-suppressive agent at start of study treatment. Note: Topical applications (e.g., rash), inhaled sprays (e.g., obstructive airways diseases), eye drops or local injections (e.g., intra-articular) and the use of systemic steroids up to a prednisone equivalent of 10 mg daily are allowed.
20. Patient has consumed Seville oranges, grapefruit, grapefruit hybrids, pomelos and exotic citrus fruits (as well as their juices) during the last 7 days prior to start of treatment. Regular orange juice is permitted.
21. Second malignancy within the past 3 years except:

    1. Adequately treated basal cell or squamous cell skin cancer (adequate wound healing is required prior to entry in the study)
    2. Adequately treated carcinoma in situ of the cervix,
    3. Prostate Cancer not requiring systemic treatment or under anti-hormonal treatment and PSA-level below upper level of normal range.
    4. Ductal breast carcinoma in situ with full surgical resection (i.e., negative margins),
    5. solid tumor treated curatively, and without evidence of recurrence for at least 3 years prior to study entry
    6. Similar condition with an expectation of > 95 % 5-year disease free survival
22. Patients with any of the following laboratory values at Screening/Baseline.

    1. Absolute neutrophil count (ANC) <1,000/mm3 [1.0 x 109/L] without Growth factor support in the last 7 days
    2. Platelets ≤ 50000/mm3 [50 x 109/L] ; patients with platelets 75000- 50000/ mm3 are eligible if thrombocytopenia is confirmed as related to myeloma bone marrow infiltration and pt. is able to receive thrombocyte concentrates
    3. Hemoglobin < 8.0 g/ dl (unless confirmed related to myeloma bone marrow infiltration and pt. able to receive blood transfusions)
    4. Serum creatinine >2 x ULN or calculated or directly measured CrCl ≤ 45 ml/min; patients with creatinin-clearance between 30-45 ml/min can be enrolled with approval by the coordinating investigator.
23. Clinically significant autoimmune haemolytic anaemia with positive Coombs test or immune thrombocytopenia
24. Patient is a woman of child-bearing potential, UNLESS they are using a double barrier method for birth control throughout the trial.

    1. Hormonal contraceptives may be affected by cytochrome P450 interactions, and are therefore considered neither indicated nor effective.
    2. Adequate barrier methods of contraception include: diaphragm, condom (by the partner), intrauterine device (copper), sponge or spermicide.
    3. Reliable contraception has to be maintained throughout the study and for 12 weeks after study drug discontinuation.
    4. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential
25. Sexually active males unless they agree to use a condom during intercourse while taking the drug. This practice should be continued for another 12 weeks after stopping treatment. Also they should not father a child during the study period or the 12 weeks post study time.

    A condom is also required to be used by vasectomized men in order to prevent delivery of the drug via seminal fluid;
26. Medical, psychiatric, cognitive or other conditions that may compromise the patient's ability to understand the patient information, give informed consent, comply with the study protocol or complete the study.
27. Patients taking non-topical medication known to be a strong inhibitor of CYP3A4. However patients who either discontinue their treatment or switch to another medication at least three days prior to registration are eligible.
28. Participation in other clinical trials within 1 month prior to enrolment except patients for supportive care studies and vaccination studies. This does not include long-term follow-up periods without active drug treatment of previous studies during the last 6 months.
29. Patient has other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment contraindicate her participation in the clinical study (e.g. uncontrolled diabetes, chronic pancreatitis, active chronic hepatitis ).

No subject will be allowed to be enrolled in this trial more than once.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-06; Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Response is assessed by quantification of monoclonal protein in serum and urine and by immunofixation of serum and urine | response assessment is performed after each cycle of therapy (28 days)

SECONDARY OUTCOMES:
Correlation of overall survival with cytogenetic characteristics deletion 17p and translocation 4;14 | Time from start of therapy until timepoint of death will be measured for all patients up to 30 months.
MEK162 Response will be categorized according to International Myeloma Working Group (IMWG) Uniform Response Criteria | response assessment after each cycle of therapy (28 days)
To evaluate the adverse events profile of LGX818/MEK162 in this indication (with respect to all adverse events and serious adverse events) | Observation period starts with the first administration of study drug and ends 30 days after the last administration of study drug or upon start of of the subsequent therapy, whatever comes first.

OTHER OUTCOMES:
Correlation of response rates and Adverse Events rates with the cytogenetic characteristics deletion 17p and translocation 4;14 | 9 months after end of study (final data analysis)
Target inhibition will be analyzed in bone marrow biopsies by detection of BRAF/MEK inhibition using immunochemistry and whole genome sequencing. | at day 28 of the first treatment cycle and at time of progression, assessed up to 30 months
Comparative genome sequencing at start of study treatment and at timepoint of progression to investigate the potential mechanism of resistance to combined BRAF/MEK inhibition | start of study treatment and at timepoint of progression, assessed up to 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc S. Raab, PD Dr. med., Principal Investigator — Medizinische Klinik V, University Hospital Heidelberg
Locations (7):
- Germany (7):
  - Universitätsklinikum Köln, Klinik I Innere Medizin, Cologne
  - Mediz. Klinik und Poliklinik 1, Universitätsklinikum Dresden, Dresden
  - Universitätsklinikum Frankfurt, Medizinische Klinik II, Frankfurt am Main
  - University Hospital Heidelberg, Med. Klinik V, Heidelberg
  - Universitätsklinikum Münster, Med. Klinik und Poliklinik A, Münster
  - Universitätsklinikum Tübingen, Medizinische Klinik II, Tübingen
  - Universitätsklinikum Würzburg, Medizinische Klinik und Poliklinik II, Würzburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Giesen N, Chatterjee M, Scheid C, Poos AM, Besemer B, Miah K, Benner A, Becker N, Moehler T, Metzler I, Khandanpour C, Seidel-Glaetzer A, Trautmann-Grill K, Kortum KM, Muller-Tidow C, Mechtersheimer G, Goeppert B, Stenzinger A, Weinhold N, Goldschmidt H, Weisel K, Raab MS. A phase 2 clinical trial of combined BRAF/MEK inhibition for BRAFV600E-mutated multiple myeloma. Blood. 2023 Apr 6;141(14):1685-1690. doi: 10.1182/blood.2022017789. PMID 36608320